CLINICAL TRIAL: NCT00812578
Title: Metabolic Effects of Vitamin D in Patients With Type 2 Diabetes - a Randomized Controlled Trial
Brief Title: Metabolic Effects of Vitamin D in Patients With Type 2 Diabetes
Acronym: ProjectD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Regionshospitalet Silkeborg (Other)
Responsible Party: MD, Med. Sci. Lotte Oerskov, Medical Department, Silkeborg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UKO-1006-2008
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-07

CONDITIONS: Type 2 Diabetes; Vitamin D Insufficiency
Keywords: Type 2 diabetes; Vitamin D insufficiency; Insulin secretion; Insulin sensitivity; Pulsatility
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cholecalciferol (Active Comparator)
  Interventions: Drug: Cholecalciferol
- Placebo pill (Placebo Comparator)
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — 8 tablets equivalent to 280 micrograms for 2 weeks and 4 tablets equivalent to 140 micrograms for 10 weeks

SUMMARY:
The purpose of the study is to examine the effect on metabolic parameters after 12 weeks of treatment with high dose vitamin D in patients with type 2 diabetes and vitamin D insufficiency.

DETAILED DESCRIPTION:
There is increasing evidence that vitamin D affects the risk of diabetes. The role of vitamin D in type 2 diabetes is suggested by cross sectional studies, where an inverse association between vitamin D status and the development of type 2 diabetes has been found. Moreover supplementation with calcium and vitamin D may attenuate increases in glycemia and insulin resistance in healthy older adults with IFG. However further research is needed to confirm these findings and to determine possible mechanisms of the preventive effect from vitamin D against diabetes. The aim of this study is to examine the effect on metabolic parameters such as glycemic control, lipid status, inflammatory markers, insulin resistance and insulin secretion in patients with type 2 diabetes and vitamin D insufficiency before and after a 12-week period of treatment with high doses of vitamin D.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Type 2 diabetes
* Patients of Danish extraction
* Vitamin D insufficiency (1,25OHvitD < 50 nmol/l)

Exclusion Criteria:

* Nephropathy (Urea > 12 mmol/l)
* S-calcium > 2,52 mmol/L
* Primary hyperparathyroidism
* Serious disease
* Malabsorption
* Sarcoidosis
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Insulin secretion and insulin resistance | 6 hours

SECONDARY OUTCOMES:
Glycemic control, lipid status, inflammatory markers, BMD | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Lotte Oeskov, MD, Principal Investigator — Medical Department, Silkeborg Hospital, Falkevej 1-3, 8600 Silkeborg, Denmark
Locations (1):
- Medical Research Unit, Medical Department M, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Kampmann U, Mosekilde L, Juhl C, Moller N, Christensen B, Rejnmark L, Wamberg L, Orskov L. Effects of 12 weeks high dose vitamin D3 treatment on insulin sensitivity, beta cell function, and metabolic markers in patients with type 2 diabetes and vitamin D insufficiency - a double-blind, randomized, placebo-controlled trial. Metabolism. 2014 Sep;63(9):1115-24. doi: 10.1016/j.metabol.2014.06.008. Epub 2014 Jun 19. PMID 25044176